CLINICAL TRIAL: NCT01359852
Title: An Open-Label Study to Investigate the Dosimetry of the Positron Emission Tomography Ligand for the Metabotropic Glutamate Receptor-2 (mGlu2R), [11C]JNJ-42491293, and Displacement by the mGlu2R Positive Allosteric Modulator JNJ-40411813 in Healthy Male Subjects
Brief Title: A Study of [11C]JNJ-42491293, a Possible PET Ligand for the mGlu2 Receptor, in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: VICE-PRESIDENT, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CR017848; 42491293EDI1001; 2010-022063-36
Record Dates: First submitted 2011-05-12; First posted 2011-05-25 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: JNJ-42491293; JNJ-40411813; Metabotropic glutamate subtype 2 receptor (mGlu2R); Positive allosteric modulator (PAM); positron emission tomography (PET)
MeSH Terms: interventions — 1-butyl-3-chloro-4-(4-phenyl-1-piperidinyl)-(1H)-pyridone

ARMS (1):
- 001 (Experimental): [11C] JNJ-42491293 + JNJ-40411813 Part C:[11C] JNJ-42491293 (300 to 370 MBq) will be dosed as an i.v.bolus injection. Volunteers will be pre-treated with JNJ-40411813 between 1.5 to 3 hours prior to the second and prior to the third PET scan,[11C] JNJ-42491293 + JNJ-40411813 Part D:[11C] JNJ-42491293 (300 to 370 MBq) will be dosed as an i.v. bolus injection.
  Volunteers will be treated with a single dose of up to 500 mg JNJ-40411813 prior to the second scan and will have a third scan at least 2 hours later to evaluate the rate of clearance of JNJ-40411813 from the brain,[11C] JNJ-42491293 Part A: [11C] JNJ-42491293 (300 to 370 MBq) will be dosed as an i.v. bolus injection and have a 120 minute PET scan.,[11C] JNJ-42491293 Part B:[11C] JNJ-42491293 (300 to 370 MBq) will be dosed as an i.v. bolus injection have a 90 minute PET scan and have arterial and venous blood sampling.
  Interventions: Drug: [11C] JNJ-42491293; Drug: [11C] JNJ-42491293 + JNJ-40411813

INTERVENTIONS:
Drug: [11C] JNJ-42491293 — Part B:[11C] JNJ-42491293 (300 to 370 MBq) will be dosed as an i.v. bolus injection, have a 90 minute PET scan and have arterial and venous blood sampling.
Drug: [11C] JNJ-42491293 + JNJ-40411813 — Part C:[11C] JNJ-42491293 (300 to 370 MBq) will be dosed as an i.v.bolus injection. Volunteers will be pre-treated with JNJ-40411813 between 1.5 to 3 hours prior to the second and prior to the third PET scan
Drug: [11C] JNJ-42491293 + JNJ-40411813 — Part D:[11C] JNJ-42491293 (300 to 370 MBq) will be dosed as an i.v. bolus injection.
  Volunteers will be treated with a single dose of up to 500 mg JNJ-40411813 prior to the second scan and will have a third scan at least 2 hours later to evaluate the rate of clearance of JNJ-40411813 from the brain
Drug: [11C] JNJ-42491293 — Part A: [11C] JNJ-42491293 (300 to 370 MBq) will be dosed as an i.v. bolus injection and have a 120 minute PET scan.

SUMMARY:
The purpose of this study is to evaluate [11C] JNJ-42491293 as a PET ligand in healthy adult volunteers.

DETAILED DESCRIPTION:
This is an open-label (volunteers will know the identity of assigned treatment) study in healthy adult volunteers and will consist of 4 consecutive parts, A, B, C, and D. Advancement to parts B, C, and D will occur only if the objectives of the preceding parts are met. Healthy adult volunteers will be recruited for each part of the study. This will be the first study in which 42491293 will be given to healthy adult volunteers. Part A will investigate the measurement of radiation (referred to as radiation dosimetry) of 42491293. Part B will measure the regional brain kinetics (activity) and binding properties of 42491293. Part C will assess the dose dependent blocking of 42491293 by 40411813 in brain tissues following single oral doses of 40411813. Part D will assess the 'duration of occupancy' of the metabotropic glutamate receptor-2 (mGluR2) positive allosteric modulator (PAM) site in the brain by 40411813 compared to peripheral clearance. In this study, 42491293 will be radio-labeled and evaluated as a potential positron emission tomography (PET) ligand for use in imaging studies of the brain to detect binding of 40411813, a compound being developed for treating patients with psychiatric conditions such as schizophrenia and anxiety disorders. In Parts A,B,C, and D, [11C] JNJ-42491293 (300 to 370 MBq) will be dosed as an i.v. bolus injection. During Part C and D, JNJ-40411813 (up to 500mg) will be administered orally (by mouth) 1.5 to 3 hours prior to scheduled PET scans.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 30 kg/m2, inclusive (BMI = weight/height2)
* Nonsmokers (at least 3 months before screening)
* Healthy on the basis of results from physical examination, vital signs, and 12-lead ECG, clinical laboratory tests performed at screening as determined by the Investigator (study physician)
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Healthy volunteers must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* History of or current medical illness that the Investigator considers to be clinically significant
* History of or current psychiatric or neurological illness including claustrophobia (an abnormal fear of being in narrow or enclosed spaces)
* Exposed to > 1 mSv of ionizing radiation participating as a volunteer in research studies in the year before the start of this study
* Any clinically significant Magnetic Resonance Imaging (MRI) abnormalities at screening, as determined by a neuroradiologist, which are relevant for the study (not applicable for part A)
* Metal implants (pacemakers, joint replacements, etc.) or metal splinters or heavy tattoos, which are relevant for MRI (not applicable for Part A).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Metabolism (uptake, distribution, and clearance) of [11C] JNJ-42491293 in brain (Part B) | Up to approximately 8 days
Adverse events (All Parts) | Up to approximately 8 days (Part A); Up approximately 8 days (Part B); Up to 16 days (Part C); Up to approximately 9 days (Part D)
Biodistribution of [11C] JNJ-42491293 (Part A) | Up to approximately 8 days
Radiation dosimetry of [11C] JNJ-42491293 (Part A) | Up to approximately 8 days
Peripheral metabolism of [11C] JNJ-42491293 (Part B) | Up to approximately 8 days

SECONDARY OUTCOMES:
Distribution of [11C] JNJ-42491293 in the brain by pre-treatment with single oral doses of JNJ-40411813 (Part C and Part D) | Up to approximately 16 days (Part C); Up to approximately 9 days (Part D)
Clearance rate of JNJ-40411813 from the brain (Part D) | Up to approximately 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.